CLINICAL TRIAL: NCT06218004
Title: Prospective Clinical Study of Envafolimab Combined With Chemotherapy in Neoadjuvant and Conversion Therapy for Head and Neck Squamous Cell Carcinoma
Brief Title: Envafolimab Combined With Chemotherapy in Neoadjuvant and Conversion Therapy for Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hairong Liu (Other)
Responsible Party: Sponsor-Investigator, Hairong Liu, Deputy Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023(112)
Record Dates: First submitted 2023-12-15; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Efficacy and Safety
MeSH Terms: interventions — Drug Therapy; envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Neoadjuvant treatment group (Experimental): envafolimab: 150 mg once every 1 week for 8 doses subcutaneously on day 1 Chemotherapy: nab-paclitaxel + cisplatin/carboplatin 3 cycles; Albumin paclitaxel 260 mg/m2, cisplatin 75 mg/m2 divided into 3 days, carboplatin AUC 5 applied on the first day.
  Interventions: Drug: Envafolimab combined with chemotherapy
- Group B: Conversion therapy group (Experimental): envafolimab: 150 mg once every 1 week for 8 doses subcutaneously on day 1 Chemotherapy: nab-paclitaxel + cisplatin/carboplatin 3 cycles; Albumin paclitaxel 260 mg/m2, cisplatin 75 mg/m2 divided into 3 days, carboplatin AUC 5 applied on the first day.
  Interventions: Drug: Envafolimab combined with chemotherapy

INTERVENTIONS:
Drug: Envafolimab combined with chemotherapy — envafolimab: 150 mg once every 1 week for 8 doses subcutaneously on day 1 Chemotherapy: nab-paclitaxel + cisplatin/carboplatin 3 cycles; Albumin paclitaxel 260 mg/m2, cisplatin 75 mg/m2 divided into 3 days, carboplatin AUC 5 applied on the first day.
  Other Names: Envafolimab

SUMMARY:
This study is a prospective clinical study. The purpose is to explore the efficacy and safety of Envafolimab combined with chemotherapy for neoadjuvant treatment or conversion treatment of locally advanced head and neck squamous cell carcinoma, and to observe the correlation between the immune microenvironment and the efficacy of immune checkpoint inhibitors, genetic changes and the efficacy in head and neck squamous cell carcinoma .

DETAILED DESCRIPTION:
This study is a prospective clinical study. The purpose is to explore the efficacy and safety of Envafolimab combined with chemotherapy for neoadjuvant treatment or conversion treatment of locally advanced head and neck squamous cell carcinoma, and to observe the correlation between the immune microenvironment and the efficacy of immune checkpoint inhibitors, genetic changes and the efficacy in head and neck squamous cell carcinoma .

After the patient signed the informed consent form, he was screened to meet the enrollment criteria and received envafolimab combined with chemotherapy according to the patient's condition.

For the first imaging evaluation, if surgical treatment can be performed, neoadjuvant therapy is required to be enrolled in group A, and 3 cycles of chemotherapy combined with envafolimab are given for re-imaging after treatment. The iRECIST criteria were used to evaluate and observe the ORR and PRO (University of Washington Head and Neck Tumor Quality of Life Scale 4th Edition (UW-QOL V4.0)), if the clinical status of the subjects is stable and the investigator evaluates that surgical treatment is feasible, the subjects can be treated with surgery, and the MPR and pCR rates are observed in postoperative pathology. After the operation, the next treatment plan (adjuvant therapy or observation) is decided according to the patient's pathological condition. If the patient develops PD during the treatment period, the subject should discontinue the study treatment.

If the imaging evaluation cannot be surgically treated, conversion therapy can be used to enroll in group B, and 3 cycles of chemotherapy combined with envafolimab can be given for re-imaging after treatment. The iRECIST criteria were used to evaluate and observe the ORR and PRO (University of Washington Head and Neck Tumor Quality of Life Scale 4th Edition (UW-QOL V4.0)), if the clinical status of the subjects is stable and the investigator evaluates that surgical treatment is feasible, the subjects can be treated with surgery, and the MPR and pCR rates are observed in postoperative pathology. After the operation, the next treatment plan (adjuvant therapy or observation) is decided according to the patient's pathological condition. If the patient develops PD during the follow-up period, the subject should discontinue the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score 0-2.
2. Age 18-80 years old, male or female.
3. Histologically confirmed locally advanced head and neck squamous cell carcinoma, including nasopharyngeal, oropharyngeal, laryngeal and hypopharyngeal cancers.（Group A enrollment criteria: locally advanced nasopharyngeal carcinoma T3/T4a any N. Locally advanced oropharyngeal carcinoma T3/T4a any N. Locally advanced laryngeal cancer T3/T4a any N, locally advanced hypopharyngeal cancer T3/T4a any N. Surgery is available as assessed by an otolaryngologist, but the scope of surgery is large and neoadjuvant treatment is required.Group B enrollment criteria: locally advanced nasopharyngeal carcinoma T4b any N. Locally advanced oropharyngeal carcinoma T4b any N. Locally advanced laryngeal cancer T4b any N, locally advanced hypopharyngeal cancer T4b any N. Patients who are evaluated by an otolaryngologist as unable to undergo surgery at present are treated with conversion therapy.）
4. Estimated survival ≥ 3 months.
5. Have at least one measurable lesion according to iRECIST criteria (spiral CT scan ≥ 10 mm).
6. Hematology: leukocytes ≥ 4000/μL, neutrophils ≥ 2.000/μL, hemoglobin ≥ 9 g/dL, platelets ≥ 90000/μL.
7. Liver function: ALT, AST, 1.5 times the upper limit of normal (ULN) <, total bilirubin < 1.5× ULN.
8. Renal function: serum creatinine < 1.5×ULN.
9. Patient has signed an informed notice and is willing and able to comply with the study plan's visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Known allergy to any of the drugs in the study;
2. Pregnant or lactating women;
3. Participated in other drug clinical trials within 4 weeks before the start of the study;
4. Those who have undergone major surgery within 28 days;
5. As judged by the investigator, the patient's tumor has a very high risk of affecting important blood vessels and causing fatal hemorrhage during treatment;
6. Have a history of severe bleeding, and have any bleeding events with a severity grade of 3 or above in CTCAE4.0 within 4 weeks prior to screening;
7. Patients with hypertension that cannot be well controlled by a single antihypertensive drug (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg);
8. Clinically significant (e.g., active) cardiovascular disease - such as cerebrovascular accident (6 months prior to ≤ randomization), myocardial infarction (6 months prior ≤to randomization), unstable angina pectoris, New York College of Cardiology (NYHA) grade II or above congestive heart failure, or severe arrhythmia that cannot be controlled with medication or has a potential impact on the trial treatment;
9. Arterior/venous thrombosis events within 6 months before the start of screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except for those who have recovered due to intravenous thrombosis caused by intravenous catheterization in the early stage of chemotherapy and judged by the investigator) and pulmonary embolism;
10. Renal insufficiency: urine routine proteinuria >2+, and confirmed 24-hour urine protein quantification > 1.0 g;
11. Long-term unhealed wounds or fractures with incomplete healing;
12. Those who have been treated with strong CYP3A4 inhibitors within one week before enrollment, or have been treated with strong CYP3A4 inducers within 2 weeks before participating in the study;
13. Symptomatic brain metastases (confirmed or suspected);
14. Presence of severe or uncontrolled infection;
15. Those who have a history of psychotropic drug abuse and cannot be quit or have a history of mental disorders;
16. Have a history of immunodeficiency, including a positive HIV test, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation, and have a history of autoimmune diseases.
17. Use of excessive high doses of glucocorticoids within 4 weeks.
18. Patients with previous and current objective evidence of history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc.;
19. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR（Objective response rate） | 12 months
  Proportion of patients whose tumors have shrunk to a prespecified value and are able to maintain the minimum time limit

SECONDARY OUTCOMES:
pCR | immediately after the surgery
  It is defined as the absence of residual infiltrates in the tissues after neoadjuvant therapy induction and surgical treatment, and no lesions can be detected in lymph node samples.The proportion of pathological complete response was achieved .
MPR | immediately after the surgery
  Defined as tumor regression with pathologic residual tumor ≤ 10% in neoadjuvant therapy induction and surgical treatment.The proportion of pathologic residual tumor ≤ 10% was achieved .
Safety of treatment | 12 months
  This includes the incidence of adverse events (AEs) and serious adverse events (SAEs), and the incidence of AEs/SAEs leading to treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Hairong Liu, Doctor, Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: No